CLINICAL TRIAL: NCT02157077
Title: A Phase III b, Multicenter Study of the Efficacy and Safety of Aflibercept Switch in Patients With Exudative AMD With Detachment of the Retinal Pigment Epithelium and Previously Treated With Ranibizumab Intravitreal Injection. (ARI2)
Brief Title: Aflibercept After Ranibizumab in Exudative Age-related Macular Degeneration
Acronym: ARI2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARI2; 2013-002869-19 (EudraCT Number)
Record Dates: First submitted 2014-03-02; First posted 2014-06-05 (Estimated); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Macular Degeneration; Wet Macular Degeneration; Retinal Degeneration; Retinal Diseases; Eye Diseases
Keywords: Eye diseases; Vision Impairment and Blindness; Eyes and Vision; Seniors; Neovascular Age-Related Macular Degeneration (AMD); Retinal Disease
MeSH Terms: conditions — Macular Degeneration; Wet Macular Degeneration; Retinal Degeneration; Retinal Diseases; Eye Diseases; Vision Disorders; Blindness | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aflibercept (Experimental): Patients will receive 2 mg of aflibercept by intravitreal injection every 4 weeks until week 8, followed by every 6 weeks to week 26
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Aflibercept — Intravitreal Injection
  Other Names: Eylea; BAY86-5321

SUMMARY:
The purpose of the current study is to evaluate the ability of Eylea to induce a regression of PED height on patients previously extensively treated by Lucentis.

The regimen proposed for this study is the 3 monthly injection followed by a 6 weeks interval injection until week 26.

DETAILED DESCRIPTION:
The regimen proposed for this study is the 3 monthly injection followed by a 6 weeks interval injection until week 26.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 50 years of age
* Active primary subfoveal choroidal neovascularization (CNV) lesions secondary to AMD including juxtafoveal lesions that affect the fovea evidenced by Fluorescein Angiography in the study eye
* Patient having been treated for at least 12 months with Ranibizumab (≥ 8 injections)
* Patient with a PED > 250 µm, defined by spectral domain optical coherent tomography (SD-OCT), measured at two consecutive visits before inclusion with any persisting sub retinal fluid at baseline
* Patient affiliated to a social security scheme
* Signed Informed Consent

Exclusion Criteria:

* Patient with subfoveal atrophy and/or atrophy with a diameter greater than 150µm in the subfoveal or juxtafoveal area
* Patient with a subfoveal fibrosis
* Subretinal hemorrhage that is either 50 percent or more of the total lesion area or 1 or more disc areas in size in the study eye.
* Scar, fibrosis or atrophy making up > 50% of total lesion in the study eye.
* Presence of retinal pigment epithelial tears or rips involving the macula in the study eye.
* History of any vitreous hemorrhage within 4 weeks prior to Visit 1 in the study eye.
* Presence of other causes of choroidal neovascularization, including pathologic myopia (spherical equivalent of -8 diopters or more negative, or axial length of 25mm or more), ocular histoplasmosis syndrome, angioid streaks, choroidal rupture, or multifocal choroiditis in the study eye or clinical evidence of diabetic retinopathy, diabetic macular edema or any retinal vascular disease other than AMD in either eye.
* Any history of macular hole of stage 3 and above in the study eye.
* Uncontrolled glaucoma (defined as intraocular pressure ≥25 mmHg despite treatment with antiglaucoma medication) or prior laser treatment for glaucoma in the study eye.
* Active intraocular inflammation or uveitis of scleritis or episcleritis in the study eye or ocular or periocular infection in either eye
* Presence or history of scleromalacia in the study eye.
* Aphakia or pseudophakia with absence of posterior capsule (unless it occurred as a result of a yttrium aluminum garnet (YAG) posterior capsulotomy) in the study eye.
* Previous therapeutic radiation in the study eye.
* History of corneal transplant or corneal dystrophy in the study eye.
* Significant media opacities, including cataract, in the study eye which might interfere with visual acuity, assessment of toxicity, or fundus photography.
* Any concurrent intraocular condition in the study eye (e.g. cataract) that, in the opinion of the investigator, could require either medical or surgical intervention during the 24 month study period.
* Any concurrent ocular condition in the study eye which, in the opinion of the investigator, could either increase the risk to the subject beyond what is to be expected from standard procedures of intraocular injection, or which otherwise may interfere with the injection procedure or with evaluation of efficacy or safety.
* Any systemic treatment with an investigational agent except dietary supplements or vitamins in the past 6 months prior to Day 1 for any condition.
* Any history of allergy to povidone iodine.
* Contraindications as listed
* Patient enrolled in another interventional research or not
* Patient already included in the study for the treatment of one of his eye
* Pregnant or nursing woman
* Lack of effective contraception for women of childbearing age

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in maximal height of pigment epithelium detachment (PED) at 12 weeks | Baseline and 12 weeks

SECONDARY OUTCOMES:
Change from baseline in central retinal thickness by SD OCT at 12 weeks | Baseline and 12 weeks
Change from Baseline in visual acuity at 12 weeks | Baseline and 12 weeks
Change from Baseline in volume of pigment epithelium detachment at 12 weeks | Baseline and 12 weeks
Association with genes involved in AMD history | genetic testing will be performed when all the particpitants will be recruited
Number of participants with adverse events from baseline to 32 weeks | from baseline to 32 weeks
Change from Baseline in pigment epithelium detachment height at 12 weeks | Baseline and 12 weeks
Change from baseline in central retinal thickness at 32 weeks | baseline and 32 weeks
Change from Baseline in pigment epithelium detachment height at 32 weeks | Baseline and 32 weeks
Change from Baseline in visual acuity at 32 weeks | Baseline and 32 weeks
Change from Baseline in volume of pigment epithelium detachment at 32 weeks | Baseline and 32 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eric Souied, MD, Study Director — Centre Hospitalier Intersommunal de Créteil
Locations (9):
- France (9):
  - Hôpital Pellegrin, Bordeaux
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Hôpital général de Dijon, Dijon
  - Centre d'Ophtalmologie Rabelais, Lyon
  - Cabinet Alpes Rétine, Montbonnot-Saint-Martin
  - CHR Hôtel Dieu, Nantes
  - Centre d'explorations ophtalmologiques de l'odéon, Paris
  - Hôpital des Quinze-Vingts, Paris
  - Clinique Mathilde, Rouen

REFERENCES:
- [Derived] Mouallem-Beziere A, Blanco-Garavito R, Richard F, Miere A, Jung C, Rozet JM, Souied EH. GENETICS OF LARGE PIGMENT EPITHELIAL DETACHMENTS IN NEOVASCULAR AGE-RELATED MACULAR DEGENERATION. Retina. 2020 Apr;40(4):663-671. doi: 10.1097/IAE.0000000000002454. PMID 30681643